CLINICAL TRIAL: NCT04926181
Title: A Phase 2 Study of Apalutamide Plus Cetrelimab in Patients With Treatment-Emergent Small Cell Neuroendocrine Prostate Cancer
Brief Title: Apalutamide Plus Cetrelimab in Patients With Treatment-Emergent Small Cell Neuroendocrine Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Rahul Aggarwal (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21553; NCI-2021-05986 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Neuroendocrine Carcinoma; Prostate Cancer; Small Cell Carcinoma
Keywords: Immunotherapy; Androgen receptor
MeSH Terms: conditions — Small Cell Lung Carcinoma; Prostatic Neoplasms; Carcinoma, Small Cell; Bulbo-Spinal Atrophy, X-Linked | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm: Apalutamide + Cetrelimab (Experimental): Participants will be given Apalutamide tablets combined with infusions of Cetrelimab in 28-day cycles, for up maximum of two years.
  Interventions: Drug: Apalutamide; Biological: Cetrelimab

INTERVENTIONS:
Drug: Apalutamide — 240 mg once daily, for a 28 day cycle
  Other Names: Erleada; Androgen Receptor Inhibitorsv(ARI); Apalutamide Oral Tablet
Biological: Cetrelimab — 480 mg given through intravenous infusion (IV) on day 1 of every 28-day treatment cycle and administered over a 60-minute infusion
  Other Names: JNJ-63723283; Anti-PD-1 antibody cetrelimab (JNJ-63723283); CET

SUMMARY:
Despite the low androgen receptor (AR) transcriptional activity of treatment-emergent small cell neuroendocrine prostate cancer, there is persistent AR expression observed in the majority of treatment-emergent small-cell neuroendocrine prostate cancer (t-SCNC) biopsies. This indicates that epigenetic dysregulation leads to reprogramming away from an AR-driven transcriptional program. Therefore, continuation of AR blockade in the form of apalutamide may provide additive benefit compared to immune checkpoint blockade alone. The investigators hypothesize that the combination of apalutamide plus cetrelimab will achieve a clinically significant composite response rate with sufficient durability of response in mCRPC patients with evidence of treatment-emergent small cell neuroendocrine prostate cancer

DETAILED DESCRIPTION:
This is a phase 2, single arm, Simon's two-stage evaluation of the combination of apalutamide plus cetrelimab in patients with mCRPC and histologic and/or genomic evidence of treatment-emergent small cell neuroendocrine prostate cancer who have previously progressed on at least one prior androgen signaling inhibitor.

Participants may continue study treatment from the time of treatment initiation until confirmed radiographic progressive disease (PD) per PCWG3 and RECIST 1.1 criteria, unequivocal clinical progression, unacceptable toxicity, or patient withdrawal, whichever occurs first, for a maximum of 24 months.

PRIMARY OBJECTIVE:

I. To determine the composite response rate as defined by achieving one or more of the following at any time point during study treatment:

1. Decline from baseline in serum PSA of >= 50% (PSA50), confirmed by repeat measurement >= 4 weeks later and/or
2. Objective response by RECIST 1.1 criteria

SECONDARY OBJECTIVES:

I. To determine safety of the combination as determined by CTCAE version 5.0.

II. To determine the median radiographic progression-free survival by PCWG3 criteria.

III. To determine the PSA50 and decline from baseline in serum PSA of >= 90% (PSA90) response proportion achieved.

IV. To determine the median PSA progression-free survival.

V. To determine the median overall survival.

VI. To determine the objective response rate and median duration of response by RECIST 1.1 criteria.

Patients will be followed up for safety evaluations 30 days and 100 days after treatment completion. Patients will be followed for overall survival every 90 days (+/- 30 days) from last dose of study treatment, until death, withdrawal of consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed prostate adenocarcinoma at the time of diagnosis, with subsequent development of metastatic castration-resistant prostate cancer. Prostate adenocarcinoma with neuroendocrine features (e.g. positive chromogranin and/or synaptophysin expression by IHC) is allowed.
2. Evidence of disease progression (PD) by PSA and/or radiographic progression by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria at the time of study entry.
3. Prior progression on at least one androgen signaling inhibitor (e.g. abiraterone acetate, apalutamide, enzalutamide, darolutamide ). Treatment with prior androgen signaling inhibitor may have been initiated in either the castration-sensitive prostate cancer (CSPC) and/or CRPC setting.
4. Patients must be evaluable for the primary endpoint of composite response and must have either serum Prostate-specific antigen (PSA) > 2 ng/mL during screening and/or measurable disease by RECIST 1.1 criteria.
5. Participants must have clinicogenomic evidence of treatment emergent small cell neuroendocrine prostate cancer as defined by one or more of the following:

   1. Histologic evidence of small cell neuroendocrine prostate cancer on evaluation of castrate resistant prostate cancer (CRPC) tissue by centralized pathology review and/or
   2. Presence of loss-of-function mutation or deletion of Retinoblastoma (RB1) gene on a Clinical Laboratory Improvement Amendments (CLIA)-approved genomic-sequencing platform. Either monoallelic or biallelic mutations in RB1 are allowed.
6. No more than one prior line of taxane-based chemotherapy administered in the metastatic castrate resistant prostate cancer (mCRPC) setting. Chemotherapy administered in the castration-sensitive setting does not count towards this limit. Prior carboplatin is allowed and does not count as an additional line of therapy when given in conjunction with taxane.
7. Castrate level of serum testosterone at study entry (<50 ng/dL). Patients without prior bilateral orchiectomy are required to remain on Luteinizing hormone-releasing hormone (LHRH) analogue treatment for duration of study.
8. No other systemic anti-cancer therapies administered other than LHRH analogue within 14 days or, 5 half-lives, whichever is shorter, prior to initiation of study treatment. Adverse Events (AEs) related to prior anti-cancer treatment must have recovered to Grade <= 1 with the exception of any grade alopecia and Grade <= 2 neuropathy.

   a. Patients receiving apalutamide prior to study entry may continue treatment at their current apalutamide dose level without requirement for wash-out period.
9. Age >= 18 years
10. Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky performance status >= 70%)
11. Demonstrates adequate organ function as defined below:

    1. Absolute neutrophil count >= 1,500/microliter (mcL)
    2. Platelets >= 100,000/mcL
    3. Hemoglobin >= 9.0 g/dL
    4. Total bilirubin <= 1.5 x institutional upper limit of normal (ULN), unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits
    5. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) <=3 X institutional upper limit of normal (<= 5 x ULN in presence of liver metastases)
    6. Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) <=3 X institutional upper limit of normal (<= 5 x ULN in presence of liver metastases)
    7. Serum creatinine <= 1.5 x institutional upper limit of normal
12. Ability to understand a written informed consent document, and the willingness to sign it.
13. Patients must agree to use adequate contraception and to not donate sperm prior to the study, for the duration of study participation, and 5 months after last administration of study treatment. Adequate contraception includes:

    1. Patients who are sexually active should consider their female partner to be of childbearing potential if she has experienced menarche and is not postmenopausal (defined as amenorrhea > 24 consecutive months) or has not undergone successful surgical sterilization.
    2. Even participants who have undergone vasectomy should still use acceptable method of contraception.
    3. Acceptable methods of contraception include hormonal combined (estrogen + progesterone) or progesterone only given orally, injected or implanted; intrauterine device (IUD), non hormonal intrauterine systems (IUS), tubal ligation, vasectomy and complete sexual abstinence.
14. Patients must be willing to undergo metastatic tumor biopsy during Screening if no biopsy has previously been done. If no metastatic lesion is safely accessible to tumor biopsy, this requirement will be waived. Bone or soft tissue lesion is allowed, but soft tissue will be prioritized. If a patient has archival tissue obtained within 90 days of cycle 1 day 1 (C1D1) the requirement for fresh tumor biopsy will be waived.

Exclusion Criteria:

1. De novo small cell carcinoma of the prostate.
2. Has participated in a study of an investigational product and received study treatment or used an investigational device other than those specified in the protocol within 2 weeks of C1D1.
3. Hypersensitivity to cetrelimab, apalutamide, or any of its excipients.
4. Has received prior radiotherapy within 2 weeks of C1D1. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (<=2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
5. Receipt of prior cetrelimab or another immune checkpoint inhibitor targeting PD-1/PD-L1 and/or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) (e.g. pembrolizumab, nivolumab, ipilimumab). Prior treatment with sipuleucel-T is allowed.
6. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients on low dose oral weekly methotrexate are allowed. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) or treatment with drugs (e.g. methimazole, neomercazole, carbimazole, etc.) that function to decrease the generation of thyroid hormone by a hyper-functioning thyroid gland (e.g., in Graves' disease) is not considered a form of systemic treatment of an autoimmune disease.
7. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Coronavirus-2019 (COVID-19) vaccine is allowed.
8. Individuals with concurrent second malignancy requiring active treatment at study entry that could affect safety or efficacy endpoints. Non-melanoma skin cancer, non-muscle invasive bladder cancer, and other carcinomas-in-situ are allowable exceptions.
9. Cardiac condition as defined as one or more of the following:

   1. Uncontrolled supraventricular arrhythmia or ventricular arrhythmia requiring treatment
   2. New York Heart Association (NYHA) congestive heart failure class III or IV
   3. History of unstable angina, myocardial infarction, or cerebrovascular accident within 6 months prior to C1D1
   4. Uncontrolled hypertension defined as systolic BP (SBP) >= 160 mm Hg and/or diastolic BP (DBP) >= 100 mmHg. Treatment and re-screening are permitted.
10. History of seizure or pre-disposing condition (e.g. brain metastases). Medications known to lower seizure threshold must be discontinued at least 4 weeks prior to C1D1.
11. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a prednisone equivalent dose of > 10 mg daily or other form of immunosuppressive therapy within 7 days prior to first dose of study drug.
12. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial (screening not required in the absence of risk factors).
13. For participants with evidence of chronic hepatitis B virus (HBV) infection (positive hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody (HBcAb)), the HBV viral load must be undetectable at the time of study enrollment (screening not required in the absence of risk factors).
14. Chronic active hepatitis C virus (HCV) infection defined as positive viral load (screening not required in the absence of risk factors).
15. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
16. Gastrointestinal disorder affecting absorption.
17. Has an active infection requiring intravenous (IV) antibiotics within 7 days prior to C1D1.
18. Use of a prohibited concomitant medication within 7 days of C1D1. Medications known to lower seizure threshold must be discontinued at least 4 weeks prior to C1D1.
19. Major surgery within 28 days prior to C1D1. Minor procedures including biopsies, dental surgery, cataract surgery, or outpatient procedure are allowed
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Composite Response Rate
Description: The composite response rate is determined by a combination of a decline from baseline in serum PSA of >= 50%, confirmed by repeat measurement ≥ 4 weeks later (PSA50) AND a complete response (CR) or partial response (PR) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria confirmed by repeat scan ≥ 4 weeks later.
Time Frame: Up to 2 years
Population: Confirmatory data required to determine response was not collected.
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Participants With Treatment-related Adverse Events (AEs)
Description: Proportion of participants with an adverse event determined to be related to study treatment, and classified using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0)
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 2
proportion of participants | 1.00

3. Secondary Outcome: Median Radiographic Progression-free Survival (PFS)
Description: PFS is defined as the time from initiation of study treatment until radiographic progression by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria or death, whichever occurs first. Response required to determine median PFS must be confirmed by repeat measurement ≥ 4 weeks later.
Time Frame: Up to 2 years
Population: Confirmatory data required to determine response was not collected.
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Participants With a >=50% Decline in PSA
Description: Defined as the proportion of participants with a demonstrated >= 50% decline from baseline serum PSA confirmed by repeat measurement >= 4 weeks after first time point at any time during the course of the study.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 2
proportion of participants | 0.5

5. Secondary Outcome: Proportion of Participants With a >=90% Decline in PSA
Description: Defined as the proportion of participants with a demonstrated >= 90% decline from baseline serum PSA confirmed by repeat measurement >= 4 weeks after first time point at any time during the course of the study.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 2
proportion of participants | 0.5

6. Secondary Outcome: Median PSA Progression-free Survival (PFS)
Description: PSA progression-free survival is defined as the time from initiation of study treatment until PSA progression as determined by PCWG3 criteria or death, whichever occurs first. Response required to determine median PFS must be confirmed by repeat measurement ≥ 4 weeks later.
Time Frame: Up to 2 years
Population: Confirmatory data required to determine response was not collected.
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival Rate
Description: The overall survival rate is the percentage of participants still alive from date of initiation of study treatment until death from any cause or censored at time of study closure.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 2
percentage of participants | 50

8. Secondary Outcome: Objective Response Rate
Description: From initiation of study treatment until maximal percent decline from baseline in sum of longest diameter (SLD) of target lesions by RECIST 1.1 criteria, confirmed by repeat scan ≥ 4 weeks later.
Time Frame: Up to 2 years
Population: Confirmatory data required to determine response was not collected.
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 0

9. Secondary Outcome: Median Duration of Response
Description: The length of time from a confirmed response per PCWG3 criteria until progression or death, whichever comes first.
Time Frame: Up to 2 years
Population: Confirmatory data required to determine response was not collected.
Arm/Group | Single Arm: Apalutamide + Cetrelimab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Single Arm: Apalutamide + Cetrelimab
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Apalutamide + Cetrelimab (N=2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Apalutamide + Cetrelimab (N=2)
Hematuria (Renal and urinary disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract infection (Infections and infestations) | 2 (6)
Fatigue (General disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
Study was terminated and closed earlier than expected due to lack of funding. The timing of study closure and patient-related events prevented the collection of confirmatory response data needed for objective response determination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT04926181/Prot_SAP_000.pdf